CLINICAL TRIAL: NCT01623310
Title: 12-Month OL Evaluating the Safety of Intranasal Administration Fluticasone BID Using OptiNose Device in Subjects With CS With or Without Nasal Polyps
Brief Title: 12-Month OL Intranasal Fluticasone Propionate BID Using OptiNose Device
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Optinose US Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPN-FLU-CS-3203
Record Dates: First submitted 2012-06-14; First posted 2012-06-19 (Estimated); Results first posted 2018-01-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Nasal Polyps
MeSH Terms: conditions — Nasal Polyps | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OPN-375 400 μg BID (Experimental): OPN-375 400 μg BID for 12 months
  Interventions: Drug: Fluticasone Propionate

INTERVENTIONS:
Drug: Fluticasone Propionate — Using Optinose Exhalation Delivery System
  Other Names: OPN-375

SUMMARY:
This is an open-label, multicenter study designed to assess the safety of intranasal administration of 400 μg of fluticasone propionate twice a day delivered by the OptiNose device in subjects with chronic sinusitis with or without nasal polyps. The study consists of an up-to-7-day pretreatment phase followed a 12-month open-label treatment phase. The duration of each subject's participation is approximately 53 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 years and older Women must

  * be practicing an effective method of birth control (eg, prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double-barrier method [eg, condoms, diaphragm, or cervical cap with spermicidal foam, cream, or gel], or male partner sterilization) before entry and throughout the study, or
  * be surgically sterile (have had a hysterectomy or bilateral oophorectomy, or tubal ligation at least 1 year before screening) or otherwise be incapable of pregnancy, or
  * be postmenopausal (spontaneous amenorrhea for at least 1 year).
* Women of child-bearing potential must have a negative serum beta-human chorionic gonadotropin (β-hCG) pregnancy test at the screening visit
* Have either:

a history of chronic sinusitis with bilateral nasal polyposis determined by nasoendoscopy at screening visit OR a history of chronic sinusitis (without polyps) for equal to or greater than 12 weeks and currently experiencing 2 or more of the following symptoms, one of which MUST be either nasal blockage/congestion or nasal discharge (anterior and/or posterior nasal discharge):

1. nasal blockage/congestion
2. nasal discharge (anterior and/or posterior nasal discharge)
3. facial pain or pressure
4. reduction or loss of smell

   * Subjects with comorbid asthma or COPD must be stable with no exacerbations (eg, no emergency room visits, hospitalizations, or oral or parenteral steroid use)within the 3 months before the screening visit. Inhaled corticosteroid use must be limited to stable doses of no more than 1,000 μg/day of beclomethasone (or equivalent; See Attachment 1) for at least 3 months before screening with plans to continue use throughout the study.
   * Must be able to cease treatment with intranasal steroids and inhaled corticosteroids (except permitted doses listed above for asthma and COPD) at the screening visit
   * Must be able to use the OptiNose device correctly; all subjects will be required to demonstrate correct use of the placebo device at the screening visit, see Section 12.1, Visit 1, screening procedures.
   * Must be capable, in the opinion of the investigator, of providing informed consent to participate in the study. Subjects must sign an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Women who are pregnant or lactating
* Inability to have each nasal cavity examined for any reason, including nasal septum deviation
* Nasal septum perforation
* Has had more than 1 episode of epistaxis with frank bleeding in the month before the screening visit
* Have evidence of significant baseline mucosal injury, ulceration or erosion (eg, exposed cartilage, perforation) on baseline nasal examination/nasoendoscopy
* History of sinus or nasal surgery within 6 months before the screening visit
* Current, ongoing rhinitis medicamentosa (rebound rhinitis)
* Have significant oral structural abnormalities, eg, a cleft palate
* Diagnosis of cystic fibrosis
* History of Churg-Strauss syndrome or dyskinetic ciliary syndromes
* Purulent nasal infection, acute sinusitis, or upper respiratory tract infection within 2 weeks before the screening visit. Potential subjects presenting with any of these infections may be rescreened 4 weeks after symptom resolution
* Planned sinonasal surgery during the period of the study
* Allergy, hypersensitivity, or contraindication to corticosteroids or steroids
* Allergy or hypersensitivity to any excipients in study drug
* Exposure to any glucocorticoid treatment with potential for systemic effects (eg, oral, parenteral, intra-articular, or epidural steroids, high dose topical steroids) within 1 month before the screening visit; except as noted in inclusion criteria for subjects with comorbid asthma or COPD
* Have nasal candidiasis
* Have taken a potent CYP3A4 inhibitor within 14 days before the screening visit; examples of these medications can be found in Section 11.6, Concomitant Medication.
* History or current diagnosis of any form of glaucoma or ocular hypertension (ie, intraocular pressure >21 mmHg)
* History of intraocular pressure elevation on any form of steroid therapy
* History or current diagnosis of the presence (in either eye) of a cataract
* Any serious or unstable concurrent disease, psychiatric disorder, or any significant condition that, in the opinion of the investigator could confound the results of the study or could interfere with the subject's participation or compliance in the study
* A recent (within 1 year of the screening visit) clinically significant history of drug or alcohol use, abuse, or dependence that, in the opinion of the investigator could interfere with the subject's participation or compliance in the study
* Positive urine drug screen at screening visit for drugs of abuse (see Section 14.5), with the exception of prescribed medications for legitimate medical conditions
* Have participated in a previous clinical trial of OPTINOSE FLUTICASONE
* Have participated in an investigational drug clinical trial within 30 days of the screening visit
* Employees of the investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Achieve Clinical Research, Birmingham, Alabama
  - PAB Clinical Research, Brandon, Florida
  - Sneeze Wheeze and Itch Associates, Normal, Illinois
  - Professional Research Network of Kansas, Wichita, Kansas
  - Best Clinical Trials, New Orleans, Louisiana
  - PMG Research of Winston Salem, Winston-Salem, North Carolina
  - HCCA Clinical Research Solutions, Middleburg Heights, Ohio
  - Allergy and Asthma Research Group, Eugene, Oregon
  - Clinical Research Solutions, Franklin, Tennessee
  - William Blake Partners, Grapevine, Texas
  - Focus Clinical Research, Draper, Utah
  - InterMountain Ear Nose and Throat, Salt Lake City, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - Premier Clinical Research, Spokane, Washington
  - Exemplar Research, Fairmont, West Virginia
  - Allergy Asthma and Sinus Center, Greenfield, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- OPN-375 400 μg: OPN-375 400 μg BID for 12 months
Period: Overall Study
Arm/Group | OPN-375 400 μg
Started | 223
Completed | 144
Not Completed | 79
Not completed — Adverse Event | 21
Not completed — Lost to Follow-up | 18
Not completed — Lack of Efficacy | 6
Not completed — Protocol Violation | 6
Not completed — Withdrawal by Subject | 25
Not completed — Became potentially child-bearing | 1
Not completed — Diagnoses of bilateral cateracts | 1
Not completed — Investigators Discretion-Noncompliant | 1

BASELINE CHARACTERISTICS:
Arm/Group | OPN-375 400 μg
Number analyzed (Participants) | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.4 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 127
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 175
  Black/African American | 45
  Asian | 2
  Other | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 223
Use of ICS treatment for polyps in past 10 years [Count of Participants; unit: Participants] | 214
Previous polyp removal surgery via polypectomy only [Count of Participants; unit: Participants] | 11
Previous sinus surgery for polyp removal or sinus surgery [Count of Participants; unit: Participants] | 80
Sinonasal Outcome Test 22 (SNOT-22) Total Score [Mean (Standard Deviation); unit: units on a scale] — SNOT-22 is validated in large populations with chronic sinusitis with and without nasal polyps. The 22 questions are used to calculate a total score (the sum of all items) and 4 subscale scores. The 22 questions are divided among 4 subscales: Rhinologic, Ear and Facial Symptoms, Sleep Function, and Psychological Issues subscales. The total score can range from 0-110, 0 being the best and 110 being the worst.
  0: No problem
  1. Very mild problem
  2. Mild or slight problem
  3. Moderate problem
  4. Severe problem
  5. Problem as bad as it can be Population: The Safety Analysis Set included all subjects who received at least 1 dose of study drug.
  units on a scale
    Pts With Polyps: number analyzed (Participants) | 34
    Pts With Polyps | 41.9 (23.27)
    Pts Without Polyps: number analyzed (Participants) | 189
    Pts Without Polyps | 39.7 (21.72)
Lund-Mackay total score [Mean (Standard Deviation); unit: units on a scale] — Assessment of nasal cavity appearance, via nasoendoscopy, used to evaluate signs of edema, discharge, crusting, scarring/adhesions, and nasal polyps, with each sign rated on a 0 to 2 scale.
  0: None 2: Worse outcome Population: The Safety Analysis Set included all subjects who received at least 1 dose of study drug.
  units on a scale
    Pts With Polyps: number analyzed (Participants) | 34
    Pts With Polyps | 1.7 (1.51)
    Pts Without Polyps: number analyzed (Participants) | 189
    Pts Without Polyps | 1.4 (1.20)
Summed Bilateral Nasal Polyp Grading Scale Score [Mean (Standard Deviation); unit: units on a scale] — Includes Chronic Sinusitis with Nasal Polyp Patients
  In subjects with nasal polyps, polyp grading of each nasal cavity was determined by a nasal polyp grading scale score measured by nasoendoscopy.
  0: No polyps
  1. Mild polyposis: polyps not reaching below the inferior of the middle turbinate
  2. Moderate polyposis: polyps reaching below the inferior border of the middle concha, but not the inferior border of the inferior turbinate
  3. Severe polyposis: large polyps reaching below the lower inferior border of the inferior turbinate
  units on a scale | 2.8 (1.17)
Nasal Polyp Surgery Eligibility [Count of Participants; unit: Participants] — Population: The Safety Analysis Set included all subjects who received at least 1 dose of study drug.
  Participants
    Pts With Polyps: number analyzed (Participants) | 34
    Pts With Polyps | 16
    Pts Without Polyps: number analyzed (Participants) | 189
    Pts Without Polyps | 11

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Patients with at least one Adverse Events
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | OPN-375 400 μg
Number analyzed (Participants) | 223
Participants | 169

2. Secondary Outcome: Sinonasal Outcome Test 22 (SNOT-22) Total Score
Description: Change from baseline to Month 3 & Month 12 in SNOT-22 Total Score
  SNOT-22 is validated in large populations with chronic sinusitis with and without nasal polyps. The 22 questions are used to calculate a total score (the sum of all items) and 4 subscale scores. The 22 questions are divided among 4 subscales: Rhinologic, Ear and Facial Symptoms, Sleep Function, and Psychological Issues subscales. The total score can range from 0-110, 0 being the best and 110 being the worst.
  0: No problem
  1. Very mild problem
  2. Mild or slight problem
  3. Moderate problem
  4. Severe problem
  5. Problem as bad as it can be
Time Frame: Baseline, Month 3, Month 12
Population: The Safety Analysis Set included all subjects who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OPN-375 400 μg
Number analyzed (Participants) | 223
units on a scale
  Change from BL to Month 3, Pts With Polyps: number analyzed (Participants) | 32
  Change from BL to Month 3, Pts With Polyps | -16.7 (15.39)
  Change from BL to Month 3, Pts Without Polyps: number analyzed (Participants) | 159
  Change from BL to Month 3, Pts Without Polyps | -18.6 (20.06)
  Change from BL to Month 12, Pts With Polyps: number analyzed (Participants) | 24
  Change from BL to Month 12, Pts With Polyps | -21.5 (21.81)
  Change from BL to Month 12, Pts Without Polyps: number analyzed (Participants) | 120
  Change from BL to Month 12, Pts Without Polyps | -21.1 (22.96)

3. Secondary Outcome: Lund-Mackay Total Score
Description: Change from baseline to Month 3, Month 12, in Lund-Mackay Total Score
  Lund-Mackay Assessment of nasal cavity appearance, via nasoendoscopy, used to evaluate signs of edema, discharge, crusting, scarring/adhesions, and nasal polyps, with each sign rated on a 0 to 2 scale 0: None 2: Worse outcome
Time Frame: Baseline, Month 3, Month 12
Population: The Safety Analysis Set included all subjects who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OPN-375 400 μg
Number analyzed (Participants) | 223
units on a scale
  Change from BL to Month 3, Pts With Polyps: number analyzed (Participants) | 32
  Change from BL to Month 3, Pts With Polyps | -0.8 (1.35)
  Change from BL to Month 3, Pts Without Polyps: number analyzed (Participants) | 162
  Change from BL to Month 3, Pts Without Polyps | -0.8 (1.21)
  Change from BL to Month 12, Pts With Polyps: number analyzed (Participants) | 24
  Change from BL to Month 12, Pts With Polyps | -0.7 (1.63)
  Change from BL to Month 12, Pts Without Polyps: number analyzed (Participants) | 120
  Change from BL to Month 12, Pts Without Polyps | -0.8 (1.18)

4. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The PGIC took less than 1 minute to complete. Subjects answered question, "Since starting the study drug, how would you rate the change in your symptoms?" Patients may answer very much improved, much improved, minimally improved, no change, minimally worse, much worse, or very much worse. Data listed below reports the total number of patients who answered very much improved, much improved, or minimally improved at the specified time.
Time Frame: Baseline, Month 3, Month 12
Population: The Safety Analysis Set included all subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | OPN-375 400 μg
Number analyzed (Participants) | 223
Participants
  Month 3, Pts With Polyps: number analyzed (Participants) | 34
  Month 3, Pts With Polyps | 27
  Month 3, Patients Without Polyps: number analyzed (Participants) | 189
  Month 3, Patients Without Polyps | 151
  Month 12, Pts With Polyps: number analyzed (Participants) | 24
  Month 12, Pts With Polyps | 22
  Month 12, Pts Without Polyps: number analyzed (Participants) | 119
  Month 12, Pts Without Polyps | 110

5. Secondary Outcome: Summed Bilateral Nasal Polyp Grading Scale Score
Description: In subjects with nasal polyps, polyp grading of each nasal cavity was determined by a nasal polyp grading scale score measured by nasoendoscopy.
  0: No polyps
  1. Mild polyposis: polyps not reaching below the inferior of the middle turbinate
  2. Moderate polyposis: polyps reaching below the inferior border of the middle concha, but not the inferior border of the inferior turbinate
  3. Severe polyposis: large polyps reaching below the lower inferior border of the inferior turbinate
Time Frame: Baseline, Month 3, Month 12
Population: Includes Chronic Sinusitis with Nasal Polyp Patients
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OPN-375 400 μg
Number analyzed (Participants) | 34
units on a scale
  Month 3: number analyzed (Participants) | 32
  Month 3 | 2.0 (1.81)
  Month 12: number analyzed (Participants) | 24
  Month 12 | 1.3 (1.19)

6. Secondary Outcome: Nasal Polyp Surgery Eligibility
Time Frame: Baseline, Month 3, Month 12
Population: The Safety Analysis Set included all subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | OPN-375 400 μg
Number analyzed (Participants) | 223
Participants
  Month 3, Pts With Polyps: number analyzed (Participants) | 32
  Month 3, Pts With Polyps | 5
  Month 3, Patients Without Polyps: number analyzed (Participants) | 162
  Month 3, Patients Without Polyps | 2
  Month 12, Pts With Polyps: number analyzed (Participants) | 23
  Month 12, Pts With Polyps | 1
  Month 12, Pts Without Polyps: number analyzed (Participants) | 120
  Month 12, Pts Without Polyps | 3

ADVERSE EVENTS:
Groups:
- Fluticasone: 400 μg of Fluticasone Propionate Twice a Day (BID) Using a Novel Bi-Directional Device
  Fluticasone Proprionate using OptiNose Device
Arm/Group | Fluticasone
All-Cause Mortality (participants affected / at risk) | 0/223
Serious Adverse Events (participants affected / at risk) | 0/223
Other Adverse Events (participants affected / at risk) | 169/223
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone (N=223)
Acute Sinusitis (Infections and infestations) | 31
Upper Respiratory Tract Infection (Infections and infestations) | 17
Bronchitis (Infections and infestations) | 6
Influenza (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 5
Intraocular Pressure Increase (Investigations) | 5
Headache (Nervous system disorders) | 21
Spontaneously Reported Epistaxis (Respiratory, thoracic and mediastinal disorders) | 25
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 39
Nasal Septum Disorder (Respiratory, thoracic and mediastinal disorders) | 32
Nasal Septum Ulceration (Respiratory, thoracic and mediastinal disorders) | 25
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis Identified via Nasal Endoscopy (Respiratory, thoracic and mediastinal disorders) | 37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreement is described in the CTA between sponsor and PI